CLINICAL TRIAL: NCT02068222
Title: An Open-Label Pilot Study to Evaluate the Antiviral Activity, Safety, Tolerability, and Pharmacokinetics of ABT-450 With Ritonavir (ABT-450/r) Dosed in Combination With ABT-530, With and Without Ribavirin (RBV) in Treatment-Naïve Subjects With Genotype 3 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Study to Evaluate the Safety and Antiviral Effect of ABT-450/Ritonavir and ABT-530 Coadministered With and Without Ribavirin in Adults With Genotype 3 Hepatitis C (HCV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-213
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Chronic Hepatitis C; Hepatitis C Virus
Keywords: Hepatitis C; HCV; Interferon Free; Chronic Hepatitis C; Hepatitis C virus; Hepatitis C Genotype 3
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — paritaprevir; pibrentasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABT-450/r and ABT-530 plus RBV (Experimental): ABT-450/r (150 mg/100 mg) once daily (QD) co-administered with ABT-530 (120 mg) once daily (QD) plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks.
  Interventions: Drug: ABT-450/ritonavir (r); Drug: ABT-530; Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: ABT-450/ritonavir (r) — Tablet
  Other Names: ABT-450 also known as paritaprevir
Drug: ABT-530 — Tablet
  Other Names: pibrentasvir
Drug: Ribavirin (RBV) — Tablet

SUMMARY:
The purpose of this study is to evaluate the safety and antiviral effect of ABT-450/r and ABT-530 coadministered with and without Ribavirin in adults with genotype 3 HCV infection.

DETAILED DESCRIPTION:
Once the efficacy and safety data were obtained from participants administered ABT-450/r + ABT-530 + RBV weight-based (Arm 1) in Study M14-213, the decision was made to end this study before subjects were enrolled into Arm 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (of non-child bearing potential) between 18 and 70 years of age with Body Mass Index ≥18 to <38 kg/m2.
* Chronic HCV genotype 3 infection prior to study enrollment and has never received antiviral treatment for HCV.
* Subject has plasma HCV RNA level > 10,000 IU/mL at Screening.
* Sexually active males must be sterile, have male partners only, or agree to use two effective forms of birth control for 7 months after stopping study drug.

Exclusion Criteria:

* History of severe, life-threatening or other significant sensitivity to any drug.
* Positive test result for Hepatitis B surface antigen (HBsAg) or anti-Human Immunodeficiency virus antibody (HIV Ab).
* Prior therapy for the treatment of HCV.
* Any current or past clinical evidence of cirrhosis.
* Any cause of liver disease other than chronic HCV-infection.
* HCV genotype co-infection with any other HCV genotype.
* Use of contraindicated medications within 2 weeks or 10 half-lives of dosing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armen Asatryan, MD, Study Director — AbbVie

REFERENCES:
- [Result] Poordad F, Landis CS, Asatryan A, Jackson DF 3rd, Ng TI, Fu B, Lin CW, Yao B, Kort J. High antiviral activity of NS5A inhibitor ABT-530 with paritaprevir/ritonavir and ribavirin against hepatitis C virus genotype 3 infection. Liver Int. 2016 Aug;36(8):1125-32. doi: 10.1111/liv.13067. Epub 2016 Feb 3. PMID 26778412

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-450/r and ABT-530 Plus RBV
Started | 10
Completed | 9
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | ABT-450/r and ABT-530 Plus RBV
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Achieve 12-week Sustained Virologic Response (SVR12)
Description: SVR12 defined as hepatitis C (HCV) ribonucleic acid (RNA) less than the lower limit of quantification (LLOQ) 12 weeks after the last actual dose of study drug.
Time Frame: 12 weeks after last dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r and ABT-530 Plus RBV
Number analyzed (Participants) | 10
percentage of participants | 90 [55.5 to 99.7]

2. Secondary Outcome: The Percentage of Subjects Who Achieve 24-week Sustained Virologic Response (SVR24)
Description: SVR24 defined as HCV RNA LLOQ 24 weeks after last dose of study drug.
Time Frame: 24 weeks after last dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r and ABT-530 Plus RBV
Number analyzed (Participants) | 10
percentage of participants | 90 [55.5 to 99.7]

3. Secondary Outcome: The Percentage of Subjects With Virologic Failure During Treatment
Description: Percentage of subjects with quantifiable HCV RNA throughout the entire treatment period, confirmed quantifiable HCV RNA after previously having unquantifiable HCV RNA, or a confirmed increase of at least one log10 in HCV RNA during treatment.
Time Frame: Up to Treatment Week 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r and ABT-530 Plus RBV
Number analyzed (Participants) | 10
percentage of participants | 10 [0.3 to 44.5]

4. Secondary Outcome: The Percentage of Subjects With Post-Treatment Relapse
Description: Percentage of subjects with confirmed quantifiable HCV RNA within 12 weeks of last dose among subjects with unquantifiable hepatitis C virus ribonucleic acid at the end of treatment.
Time Frame: Within 12 weeks after the last dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-450/r and ABT-530 Plus RBV
Number analyzed (Participants) | 9
percentage of participants | 0 [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 16.5 weeks); serious adverse events (SAEs) were collected from the time informed consent was obtained through end of study (up to 41 weeks).
Description: Treatment-emergent adverse events are defined as any adverse event (AE) with an onset date that is after the first dose of study drug and no more than 30 days after the last dose of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Groups:
- ABT-450/r and ABT-530 Plus RBV: ABT-450/r (150 mg/100 mg) once daily (QD) co-administered with ABT-530 (120 mg) QD plus weight-based RBV (dosed 1,000 or 1,200 mg daily divided twice a day) for 12 weeks.
Arm/Group | ABT-450/r and ABT-530 Plus RBV
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-450/r and ABT-530 Plus RBV (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 1
DRY EYE (Eye disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
FAECES SOFT (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 2
CHEST DISCOMFORT (General disorders) | 1
FATIGUE (General disorders) | 4
MALAISE (General disorders) | 1
PAIN (General disorders) | 1
PYREXIA (General disorders) | 1
THIRST (General disorders) | 1
ACARODERMATITIS (Infections and infestations) | 1
ORAL HERPES (Infections and infestations) | 1
RHINITIS (Infections and infestations) | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 1
HAEMOGLOBIN DECREASED (Investigations) | 1
ABNORMAL LOSS OF WEIGHT (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
BALANCE DISORDER (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 1
IRRITABILITY (Psychiatric disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.